CLINICAL TRIAL: NCT03540433
Title: Evaluation of POCD-Census Prospective, International Observation Study
Brief Title: International Observational Study on Perioperative Cognitive Trajectories (POCD Census International/PCI)
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Claudia Spies, Head of the Department of Anesthesiology and Intensive Care Medicine (CCM/CVK), Charite University, Berlin, Germany
Other Study IDs: PCI
Record Dates: First submitted 2018-05-17; First posted 2018-05-30 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Postoperative Cognitive Deficit (POCD); Neurocognitive Disorders
MeSH Terms: conditions — Neurocognitive Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: Surgical patients aged ≥70 years
- Control group: Healthy subjects, aged ≥70 years, American Society of Anesthesiologists (ASA) I+II+III, no surgery

SUMMARY:
The purpose of this international, multi-centre observational study is to describe perioperative cognitive changes (pre-existing neurocognitive disorder [NCD], postoperative delirium [POD] and Postoperative Cognitive Dysfunction [POCD]) up to five years after elective surgery in a mixed cohort. Measurements and definitions of cognitive outcomes will be based on current consensus and used for further harmonization in future clinical studies on perioperative cognitive trajectories. This is a feasibility approach to identify an effective screening procedure and estimate loss to follow up rates for the planning of future intervention studies. Data from this trial may also serve to facilitate and implement time effective cognitive screening and risk stratification concerning postoperative cognitive decline in the anaesthesiological preoperative assessment.

DETAILED DESCRIPTION:
This international observational study on perioperative cognitive trajectories (POCD census international/PCI) has been designed as a pilot study to allow a peer reviewed process of four international test centres on measurement of perioperative acute and long-term cognitive outcome. Data from standard clinical treatment of 500 patients age ≥ 70 years scheduled for elective surgery (stratified according to preoperative assessment of frailty and monitored by intraoperative depth of anaesthesia) will be supplemented by guideline conform delirium- analgesia- and sedation screening until day 5 after surgery, I-Pad based neuropsychological testing [Cambridge Neuropsychological Test Automated Battery - CANTAB connect] pre-operatively, 3 months, 1- 2- and 5 years after surgery, a paper-based verbal fluency test (animal naming test from Addenbrooke's Cognitive Examination Revised (ACE-R)), a paper based test on executive function (Trailmaking Test), cognitive screening tests (Montreal Cognitive Assessment (MOCA) and Mini-Cog), and concomitant questionnaires to assess functional status, self- and by proxy rating of cognitive performance, psychological factors (depression, perioperative anxiety, stress, resilience and coping), social support, perioperative anxiety, stress, resilience and coping, as well as risk consumption of alcohol and tobacco.

A non-surgical control group of 100 study participants who are not scheduled for surgery will be followed up at the same time points as the surgical cohort for scaling of cognitive data and definition of cut off values to define significant cognitive decline.

Secondary outcome measures of this trial comprise levels and changes in molecular biomarkers involved in Alzheimer's dementia etiology sampled from spinal fluid on induction of spinal anaesthesia and sampled from blood in all patients.

Retrospective comparison collective (01/01/2017 to 01/01/2022):

A group of around 8000 surgical patients aged 65 and older at the Charité will be examined as control group. This control group is required for various questions, especially influencing factors with regard to the postoperative outcome of delirium, and aims to test the predictive ability of clinical routine data with regard to postoperative delirium. As part of the multimodality of this retrospective comparative cohort study, in cooperation with PD. Dr Scheel and in collaboration with Prof. Dr. Finke, cranial MRI scans analyzing routine data from the Institute of Neuroradiology. The subject of the investigation is initially the entire electronic routine data of the control group, including the existing cranial MRI scans.

ELIGIBILITY:
Inclusion Criteria:

* Surgical patients at Campus Virchow- Klinikum and Campus Charité Mitte
* Aged ≥ 70 years
* Informed consent

Exclusion Criteria:

* Manifest dementia
* Lack of willingness to store and disseminate pseudonymized disease data as part of the clinical trial
* Lack of readiness to participate in the follow-up examinations and contact to make an appointment
* Placement in an institute under judicial or official orders (according to German drug Law §40 (1) 4)
* Persons without a permanent residence or other circumstances that call into question the availability by telephone or post for postoperative examination
* Employees of the respective study centers
* illiteracy
* Patients with a neuropsychiatric condition that limits the performance of neurocognitive testing
* Patients with hearing and / or vision problems that limit the performance of neuro-cognitive testing
* Simultaneous participation in a prospective clinical intervention study (apart from the desired parallel participation in the anaesthesiological study Praep-Go, EA1/225/19)

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Surgical patients aged ≥70 years
Sampling Method: Probability Sample
Enrollment: 173 (Actual)
Dates: Start 2018-06-08 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative cognitive dysfunction (POCD) | Up to 1 year
  Neuropsychological testing

SECONDARY OUTCOMES:
Incidence of postoperative cognitive dysfunction (POCD) | Up to 5 years
  Neuropsychological testing
Positive cognitive screening | Up to 5 years
  Short neuropsychological testing
Mild Neurocognitive Disorder | Up to five years
  Definition according to DSM-V as proposed in Evered L et al. Recommendations for the nomenclature of cognitive change associated with anaesthesia and surgery. Br J Anaesth, Anesthesiology, Can J Anesth, Anesth Analg, J Alz Dis, acta scandinavica anaesthesiologica (Joint Publication) 2017; Accepted, In Press. We will use an I-pad based neuropsychological test battery (CANTAB connect), and cognitive screening instruments (MOCA, Mini-Cog™ and Animal naming test on verbal fluency from ACE-R) for assessment of cognitive function, MMQ and IQ-code for self- or by proxy reported cognitive concern and ADL/IADL for assessment of functional status. Mild/major Neurocognitive Disorder measured at baseline (pre-existing NCD) 3 months and 1 year (with specifier 'POCD'), 2- and 5 years after surgery
Major Neurocognitive Disorder | Up to five years
  Definition according to DSM-V as proposed in Evered L et al. Recommendations for the nomenclature of cognitive change associated with anaesthesia and surgery. Br J Anaesth, Anesthesiology, Can J Anesth, Anesth Analg, J Alz Dis, acta scandinavica anaesthesiologica (Joint Publication) 2017; Accepted, In Press. We will use an I-pad based neuropsychological test battery (CANTAB connect), and cognitive screening instruments (MOCA, Mini-Cog™ and Animal naming test on verbal fluency from ACE-R) for assessment of cognitive function, MMQ and IQ-code for self- or by proxy reported cognitive concern and ADL/IADL for assessment of functional status. Mild/major Neurocognitive Disorder measured at baseline (pre-existing NCD) 3 months and 1 year (with specifier 'POCD'), 2- and 5 years after surgery
Cerobrospinal fluid biomarker for diagnosing dementia | Up to five years
  Patients for spinal anesthesia who consented on lumbar puncture receive biomarkers analysis from spinal fluid (beta Amyloid 1-40, beta-Amyloid 1-42, beta-Amyloid Ratio (42/40*10), phospho-TAU, Protein 14-3-3, PRPSc, TAU (Gesamt-Tau)).
Blood biomarker for diagnosing dementia | Up to five years
  Patients consented on blood sampling receive biomarker analysis from blood (Apolipoprotein E).
Findings of memory consultation session | Up to five years
Comorbidities | Up to five years
  Comorbidities will be quantified by use of Charlson Comorbidity index
Nutritional status | Up to five years
  Changes in the nutritional status after elective surgery are measured by a questionnaire.
Malnutrition 1 | Up to five years
  Malnutrition is measured by the Body mass index
Malnutrition 2 | Up to five years
  Malnutrition is measured by weight
Malnutrition 3 | Up to five years
  Malnutrition is measured by weight
Dental health | Up to five years
  The dental status is determined by tooth doctors
Sarcopenia | Up to five years
  The composite outcome measure "Sarcopenia" is defined by the following three criteria: 1) low muscle strength (hand grip strength), 2) low muscle quantity (calf circumference and 3) low physical performance (gait speed). Criterion (1) identifies probable sarcopenia, additional documentation of criterion (2) confirms sarcopenia diagnosis, and if all criteria (1), (2) and (3) are met, sarcopenia is considered severe.
Calf circumference | Up to five years
  Calf circumference is measured in a standardized position and documented in centimeter.
Arm circumference | Up to five years
  Arm circumference is measured in a standardized position and documented in centimeter.
Adherence to Mediterranean diet (MD) | Up to five years
  Adherence to Mediterranean diet (MD) is measured with a German Mediscore, could range from 0 to 9, with higher scores (6-9) indicating greater MD adherence.
Nutrition in the hospital | Up to five years
  Participants will be followed for the duration of hospital stay, an expected average of 7 days
Physical activity | At the beginning of the observation
  Physical activity is evaluated by interviewing the Patient.
Surgical risk | Participants will be followed up during surgery, an estimated duration of 1 hour
  Surgical risk will be described by type and length of surgery and perioperative cardiac risk estimation as described in Anästh Intensivmed 2017; 58:349-364.
Anaesthesiological Risk 1 | At the beginning of the observation
  Anaesthesiological risk will be described by American Society of Anesthesiologists Classification (ASA Class)
Anaesthesiological Risk 2 | Participants will be followed up during surgery, an estimated duration of 1 hour
  Anaesthesiological risk will be measured by length of anesthesia
Anaesthesiological Risk 3 | Participants will be followed up during surgery, an estimated duration of 1 hour
  Anaesthesiological risk will be measured by type of anaesthesia
Intraoperative depth of anaesthesia | Participants will be followed up during surgery, an estimated duration of 1 hour
  Intraoperative depth of sedation will be monitored with changes in the pattern and power spectrum of EEG-raw data measured with the Masimo SedLine® brain function monitoring for Root®, Narcotrend®, BIS™ and additionally quantified by indices [e.g. PSI or BIS-index] and burst suppression ratio.
Depth of sedation on the Intensive Care Unit | Participants will be followed for the duration of intensive care unit stay, an expected average of 5 days
  Sedation is measured by Richmond Agitation Sedation Scale.
Sedation on the peripheral ward | Participants will be followed for the duration of hospital stay, an expected average of 7 days
  Sedation is measured by Richmond Agitation Sedation Scale.
Agitation on the peripheral ward | Participants will be followed for the duration of hospital stay, an expected average of 7 days
  Agitation describes a clinical state in which the patient may be impulsive and attempt to get out of bed, to wander, and to fall (which may lead to further injury or death) and attempt to remove IV lines, tubes, or catheters.
Incidence of postoperative delirium | Up to 5 days
  Postoperative delirium rate, defined according to Diagnostic and Statistical Manual of Mental Disorders (DSM-V), CAM/CAM-ICU, Nu-DESC and Chart Review.
Severity of postoperative delirium | Up to 5 days
  Postoperative delirium rate, defined according to Confusion assessment method - severity(CAM-S); Delirium Rating Scale Revised (DSR-R-98), Intensive Care Delirium Screening Checklist (ICDSC) and Nursing Delirium Screening Scale (Nu-DESC).
Duration of Delirium | Participants will be followed for the duration of hospital stay, an expected average of 7 days
  Duration of postoperative delirium, defined according to medical evaluation, measured in days
Pain scale for patients able of pain self-assessment | Up to hospital discharge, an expected average of 5 days
  Pain during hospital stay will be measured with the Numeric Rating Scale (NRS-V).
Pain scales for patients unable of pain self-assessment | Up to hospital discharge, an expected average of 5 days
  For patients unable of pain self-assessment (e.g. ventilated patients, patients in delirious state or patients with stroke affecting language skills) observer-rated pain scales will be applied: Behavioural Pain Scale (BPS for ventilated) and BPS-NI (for non-ventilated) patients, Critical-Care Pain Observation Tool (CPOT) during hospital stay.
Intensive care unit length of stay | Participants will be followed for the duration of intensive care unit stay, an expected average of 5 days
  Intensive care unit length of stay describes every day spent in an ICU bed.
Hospital length of stay | Participants will be followed for the duration of hospital stay, an expected average of 7 days
  Hospital length of stay describes every day spent in an hospital.
Perioperative Anxiety | Up to 5 days
  Perioperative anxiety will be measured with APAIS preoperatively and the Faces Anxiety Scale (FAS) and during hospital stay.
Perception of stress | Up to 5 days
  Stress is measured by Perceived Stress Questionnaire 20
Stress level | Up to 5 days
  Stress level is measured by stress thermometer
Generalized anxiety | Up to 5 days
  Anxiety will be measured with the Generalized Anxiety Disorder 7-Item Scale (GAD-7)
Depression | Up to 5 years
  Depression is measured by PHQ-8. Scores represent:0-5 = mild, 6-10 = moderate, 11-15 = moderately severe, 16-20 = severe depression
Quality of sleep | Up to 5 years
  Quality of sleep is measured by the Insomnia Severity Index.
Routine laboratory | Up to hospital discharge, an expected average of 7 days
Organ dysfunctions | Up to hospital discharge, an expected average of 7 days
  Organ dysfunctions are evaluated according to the Clavien-Dindo classification of surgical complications
Subjective/By proxy assessment of cognitive impairment | Up to five years
Medication | Up to 5 years
  Prescribed regular drug intake from baseline at all follow ups including perioperative application of drugs, infusions and transfusions will be evaluated.
Quality of life | Up to 5 years
  Quality of life will be measured with the EQ-5D-5L
Level of dependency | Up to 5 years
  Level of dependency will be measured with with ADL/IADL, single items concerning patients' living situation and the BSSS-17 (Berlin Social Support Scales).
Plausibility check variables | Up to 5 years
  Variables affecting performance of cognitive testings
Re-admission | Up to 5 years
  Hospital readmission is an episode when a patient who had been discharged from a hospital is admitted again within a specified time interval.
Revison surgery | Up to 5 years
  Surgery performed to replace or compensate for a failed implant or to correct undesirable sequelae of previous surgery.
Outpatient treatment | Up to 5 years
  Treatment outside of the hospital in an associated facility for diagnosis or treatment.
Mortality | Up to 5 years
  The number of deaths in a given period.
Dementia | Up to 5 years
  Dementia reported as clinical diagnosis based on DSM-5 criteria for major NCD either through neuropsychological evaluation at a memory clinic or as a research diagnosis based on neuropsychological test values (CANTAB/MOCA), cognitive concern (MMQ/IQCODE) and functionality (ADL/IADL).
Motivational incongruence | Up to five years
  The incongruence questionnaire (Der Inkongruenzfragebogen)
Leisure behavior | Up to five years
  Questionnaire on frequency of cognitively stimulating leisure activities
Demographic variables | Up to five years
Living conditions | Up to five years
Postoperative electroencephalography (EEG) spectral analysis with band power | Up to seven days
  Spectral analysis with band power are measured by EEG at third postoperative day and delirium dependent until postoperative day 7.
Evaluation of pain | Up to three months
  Pain is measured with dolosys paintracker
Loneliness | Up to five years
  Loneliness is measured with the UCLA-Loneliness-Scale (3 items)
Social support | Up to five years
  Social support is measured with the Berliner Social-Support Skalen BSSS-17
Living situation | Up to five years
  Living situation is measured with te question: How do you live?

OTHER OUTCOMES:
Obesity 1 | At the beginning of the observation
  Obesity is measured by body mass index (BMI)
Obesity 2 | At the beginning of the observation
  Obesity is measured by waist to hip ratio
Variables of adjusting | At the beginning of the observation
  Reading / writing weakness, hendedness, native speaker
Frailty | At the beginning of the observation
  Frailty will be measured by Fried's criteria (Physical Frailty Phenotype), Fried et al: Frailty in older adults: evidence for a phenotype. J.Gerontol.A Biol.Sci.Med.Sci. 2001; 56: M146-M156 and evaluated in a short comprehensive geriatric assessment as decribed by Birkelbach, O. et al. Warum und wie sollte ich Frailty erfassen? - ein Ansatz für die Anästhesieambulanz. Anasthesiol. Intensivmed. Notfallmedizin Schmerztherapie 52, 765-776 (2017).
Cognitive Reserve | At the beginning of the observation
  Level of education (years of formal training, last occupation, ISCED-2011 and crystalline intelligence [IQ-variable calculated with NART/MWT-A or other national equivalent ] will be used to evaluate cognitive reserve.
Crystalline Intelligence | At the beginning of the observation
  Mehrfachwahl-Wortschatz-Intelligenztest (MWT-A) and National Adult Reading Test (NART)
Previous professional activity | At the beginning of the observation
  Interview guide employment situation and previous professional activity adapted to Engstler (2017); Classification according to ISCO 08; Workload indices according to Kroll (2011)
Delusion proneness | At the beginning of the observation
  Delusion proneness is measured by Peter's Delusion Inventory
Physical activity | At the beginning of the observation
  History of physical activity less than 30 minutes / day (i.e. moderate increase in heart rate due to fast walking, cycling or other exercise)
Pre-operative electroencephalography (EEG) spectral analysis with band power | At the beginning of the observation
  Spectral analysis with band power are measured by EEG
Preoperative Cognitive Impairment (PreCI) | At the beginning of the observation
  Preoperative Cognitive Impairment (PreCI) is measured by computerized and paper pencil tests

CONTACTS AND LOCATIONS:
Locations (3):
- Germany (3):
  - Arbeitsbereich Physikalische Medizin, Berlin
  - Internistische Hausarztpraxis, Berlin
  - Department of Anesthesiology and Intensive Care Medicine Berlin (CCM/CVK), Charité - Universitätsmedizin Berlin, Berlin

IPD SHARING:
Plan to Share IPD: No